CLINICAL TRIAL: NCT05625919
Title: A Phase Ⅰb/Ⅱ Multi-center Study of Safety and Efficacy of Sirolimus for Injection (Albumin-bound) in Patients With Advanced Malignant Perivascular Epithelioid Cell Tumor (PEComa)
Brief Title: A Study of Safety and Efficacy of Sirolimus for Injection (Albumin-bound) in Patients With Advanced Malignant Perivascular Epithelioid Cell Tumor (PEComa)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-004
Record Dates: First submitted 2022-11-14; First posted 2022-11-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignant Perivascular Epithelioid Cell Tumor (PEComa)
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms | interventions — Sirolimus; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus for Injection (Albumin-bound) (Experimental): Sirolimus for injection (Albumin-bound) will be administered intravenously on day 1and day 8 every 21 days (a cycle).
  Interventions: Drug: Sirolimus for Injection (Albumin Bound)

INTERVENTIONS:
Drug: Sirolimus for Injection (Albumin Bound) — Sirolimus for injection (Albumin-bound), intravenously, once a week, 21 days per cycle (two weeks-on and one week-off)

SUMMARY:
This is a phase Ⅰb/Ⅱ multi-center study of safety and efficacy of Sirolimus for Injection (Albumin-bound) in patients with advanced malignant perivascular epithelioid cell tumor (PEComa).

DETAILED DESCRIPTION:
This is a non-randomized, multi-center, open-label, Phase Ⅰb/Ⅱ clinical trial. For phase Ⅰb, patients must have a histologically confirmed diagnosis of advanced soft tissue sarcomas (including malignant PEComa, accounting for at least 1/2) that have failed standard treatment (disease progression or relapse or intolerance, such as chemotherapy, radiotherapy, targeted therapy, etc.) or lack effective treatment. The recommended phase II dose (RP2D) will be determined in phase Ⅰb. For phase Ⅱ, patients must have a histologically confirmed diagnosis of malignant PEComa that is either metastatic or locally advanced and for which surgery is not a recommended option. Phase Ⅱ will use the recommended dose and dosing regimen from Phase Ⅰb.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, and Phase Ⅰb: Patients with histologically confirmed diagnosis of advanced soft tissue sarcomas (including malignant PEComa, accounting for at least 1/2) have failed standard treatment (disease progression or relapse or intolerance to chemotherapy, radiotherapy, targeted therapy, etc.) or lack effective treatment; Phase Ⅱ: Patients must have a histologically confirmed diagnosis of malignant PEComa that is either metastatic or locally advanced and for which surgery is not a recommended option.

[Malignant PEComas displaying 2 or more of the features of large size (> 5 cm), infiltrative growth, high nuclear grade, cellular necrosis, mitoses ≥1/50 high power field (HPF), or vascular invasion]

* At least 1 measurable lesion as defined by RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Life expectancy >3 months.
* Patient must have the following biological parameters levels at screening (without blood transfusion, EPO, G-CSF and other medical support within14 days prior to screening tests):

Blood tests: Absolute neutrophil count (ANC) ≥1.5 × 10^9/L; Platelet count ≥100 × 10^9/L; Hemoglobin ≥90 g/L; Renal function tests: serum creatinine ≤1.5 x upper limit of normal (ULN); Liver function tests: Total bilirubin ≤1.5 x ULN (Patients with liver metastases, bile duct obstruction, or confirmed Gilbert syndrome: ≤ 3×ULN); AST and ALT ≤2.5 x ULN (≤5 x ULN if attributable to liver metastases); Blood clotting function tests: INR or PT ≤ 1.5 × ULN; APTT≤ 1.5 × ULN;

* Fasting serum triglycerides<300 mg/dL(3.42 mmol/L), fasting serum cholesterol < 350 mg/dL ( 9.07mmol/L; ).
* Fasting blood glucose (FPG) < 7.8 mmol/L and HbA1c < 8%.
* Women of child-bearing potential, or men whose partners are women of childbearing age must agree to use reliable contraceptive methods during the trial period and at least 6 months after the last administration; women of childbearing age must have a negative serum pregnancy test within 7 days prior to the first administration, should not be breast feeding.
* Patients must give informed consent to the study prior to the trial and voluntarily sign informed consent form.

Exclusion Criteria:

* Anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy within 4 weeks prior to the first dose of study drug, with the following special requirements:

Nitrosoureas (eg, carmustine, lomustine, etc.) or mitomycin C within 6 weeks prior to the first dose of study drug; Oral fluorouracils and small molecule targeted drugs within 2 weeks or 5 half-lives (whichever is longer) before the first dose of study drug; Traditional Chinese medicines with anti-tumor indications within 2 weeks prior to the first dose of study drug;

* Received other unmarketed clinical investigational drug within 4 weeks prior to the first dose of study drug.
* Major surgical procedures within 4 weeks prior to the first dose of study drug or not fully recovered from any previous invasive procedures.
* Received systemic glucocorticoids (prednisone > 10 mg/day or equivalent doses) or other immunosuppressive therapy within 2 weeks prior to the first dose of the study drug [with the following exceptions: treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of glucocorticoids for prophylaxis (eg, prevention of contrast allergy)].
* Infection that required systemic anti-infective therapy (oral or IV) within 2 weeks before enrollment.
* Inactivated or live attenuated vaccine or novel coronavirus vaccine within 30 days before the first dose.
* Use of strong inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study drug, or requiring concomitant treatment during the study.
* History of other malignancies within 5 years prior to the first dose of the study drug, except in the following cases: cured basal cell or squamous cell skin cancer, superficial bladder cancer, prostatic carcinoma in situ, carcinoma in situ of the cervix, breast carcinoma in situ, etc., or locally curable cancer that has been disease-free for 5 years;
* Liver-directed therapy is required within 2 months of enrollment. Prior treatment with radiotherapy (including radio-labeled spheres and/or cyberknife, hepatic arterial embolization (with or without chemotherapy) or cyrotherapy/ablation) is allowed if these therapies does not affect the areas of measurable disease being used for this protocol.
* History of serious cardiovascular disease, such as severe heart rhythm or conduction abnormalities (ventricular arrhythmias requiring clinical intervention, grade Ⅱ or Ш atrioventricular block, etc.). History of myocardial infarction, unstable angina, heart failure, New York College of Cardiology (NYHA) grade Ⅱ and above, and coronary artery bypass surgery within 6 months before the first dose of the study drug; Left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 msec (male) or female QTcF > 470 msec (female), etc.
* Unresolved toxicity from prior anti-tumor therapy greater than Grade 1 as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.(except for alopecia and any other toxicities that have no safety risk judged by the investigator).
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, or other evidence of uncontrollable central nervous system metastases or meningeal metastases that not eligible for inclusion determined by the investigator.
* Hydrothorax, ascites or pericardial effusion with clinical symptoms or required symptomatic treatment.
* Patients with angiomyolipoma(AML) or lymphangioleiomyomatosis (LAM).
* History of serious lung disease, such as interstitial lung disease and/or pneumonitis, or pulmonary hypertension, or pre-existing severely impaired lung function.
* Pre-existing thyroid abnormality is allowed provided thyroid function can be controlled with medication.
* Known hypersensitivity or intolerance to any ingredient in the study drug.
* History of autoimmune disease (except tuberous sclerosis), immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency disease, or history of organ transplantation.
* Active Hepatitis B or Hepatitis C, or active syphilis infection Active Hepatitis B: HBsAg-positive with HBV DNA titer ≥ 1 × 10^3 IU/mL; Patients are eligible for enrollment if they are HBsAg positive with peripheral blood HBV-DNA < 1 × 10^3 IU/mL if, in the opinion of the investigator, the patient's chronic hepatitis B is in a stable phase and does not increase the subject's risk.

Active Hepatitis C: HCV antibodies -positive with HCV RNA-positive; Active syphilis infection: Treponema pallidum antibodies (RPR or TRUST)-positive or presence of syphilis infection requiring systemic therapy.

* Severe concomitant diseases that endanger patient safety, interfere the compliance of the study procedure (such as uncontrollable hypertension, active gastrointestinal bleeding, etc.) or other reasons that make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
AE and SAE occurrence and frequency in phase Ⅰb | Up to 2 years
Dose-limiting toxicities (DLT) | Cycle 1 (Up to 21 days)
Maximum tolerated dose (MTD) | Cycle 1 (Up to 21 days)
Recommended phase 2 dose (RP2D) | Cycle 1 (Up to 21 days)
Overall response rate (ORR) in phase Ⅱ | Up to 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) in phase Ⅰb | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Overall survival (OS) | Up to 2 years
AE and SAE occurrence and frequency in phase Ⅱ | Up to 2 years
Area under the plasma concentration versus time curve (AUC) | Up to 2 years
Peak Plasma Concentration (Cmax) | Up to 2 years
Peak time (Tmax) | Up to 2 years
Terminal half-life (t½) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China